CLINICAL TRIAL: NCT05890820
Title: Evaluation of the Effect of Preoperative Nutritional Risk Parameters on Postoperative Pulmonary Complications in Geriatric Patients Who Underwent Lung Resection for Malignancy, a Prospective Observational Study
Brief Title: The Effect of Nutritional Risk Parameters on Postoperative Pulmonary Complications in Geriatric Thoracic Surgery Cases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Özgür Cirik, Associate Proffessor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: E-53610172-799-207700439
Record Dates: First submitted 2023-05-16; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer; Nutrition, Healthy; Postoperative Complications
MeSH Terms: conditions — Lung Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Preoperative nutritional assessment — Preoperative nutritional assessment and postoperative pulmonary complications

SUMMARY:
Preoperative evaluation of nutritional status in geriatric patients with lung cancer and implementation of these practices in elective patients are very important in terms of reducing postoperative complications and accelerating hospital discharge. For this purpose, many nutritional assessments and measurements are used. Our aim in this study was to evaluate the relationship between preoperative nutritional status and postoperative pulmonary complications in patients undergoing thoracic surgery for geriatric lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age
* Lung Cancer
* Patients undergoing thoracic surgery

Exclusion Criteria:

* Refusal to participate in the study
* Patients with a diagnosis of hematological malignancy
* Patients with missing data required for research

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients over 65 years of age with lung malignancy and undergoing thoracic surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
FFMI - Fat-Free Mass Index | 24 hours
  FFMI is an abbreviation for lean mass index. It defines the amount of your muscle mass relative to height and weight. The FFMI is part of the well-known and similar BMI family of body indexes. The effect of FFMI values on postoperative patient stay, intensive care unit stay, complications and postoperative mobilization time in lung cancer patients will be evaluated. Each patient will be evaluated by measuring the preoperative FFMI value 24 hours before.

SECONDARY OUTCOMES:
BMI (Body Mass Index) | 24 hours
  BMI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass. The effect of BMI values on postoperative patient stay, intensive care unit stay, complications and postoperative mobilization time in lung cancer patients will be evaluated. Each patient will be evaluated by measuring the preoperative BMI value 24 hours before.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Sanatoryum Education and Research Hospital, Ankara, Keçioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No